CLINICAL TRIAL: NCT04226573
Title: The Effect of Preoperative Anxiety on Fetal Cord Blood Tumor Necrosis Factor-Alpha and Interleukin-6 Levels in Pregnant Women
Brief Title: Effect of Preoperative Anxiety on Fetus in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Ökkeş Hakan Miniksar, Assistant Professor, Bozok University
Other Study IDs: 2019.10.231
Record Dates: First submitted 2019-12-11; First posted 2020-01-13 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Preoperative Anxiety; Cytokines
Keywords: Preoperative anxiety; Umbilical cord blood; Cytokines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low anxiety, Middle and High anxiety: State Trait Anxiety İndex Scale: Values of less than 60, Low anxiety State Trait Anxiety İndex Scale: Values above 60, Middle and High anxiety
  Interventions: Other: Preoperative anxiety levels

INTERVENTIONS:
Other: Preoperative anxiety levels — Serums were separated from blood samples taken from all patients in the study, Using the anti-human TNF-α and IL-6 enzyme-linked immunosorbent assay (ELISA) kits in the Elisa device, the TNF-α and IL-6 cytokines will be measured to determine their concentration.
  No routine blood will be drawn during the procedures. Preoperative anxiety levels will be evaluated with STAI-Continuity and STAI-Statefulness scale.
  Other Names: Tumor Necrosis Factor-Alfa and İnterleukin-6 cytokine concentrations in fetal cord blood

SUMMARY:
In the preoperative period, 60-80% of the patients had anxiety symptoms. This rate increases even more during pregnancy. There are a number of studies examining the role of anxiety symptoms on fetal outcome, but the mechanisms that explain the effects of maternal stress are not fully understood.

The most extensively studied cytokines in neuropsychiatric disorders are TNF-α and IL-6 due to their effects on the central nervous system. TNF-α levels have been reported to be elevated in anxiety disorders. In our study, the investigators aimed to determine the relationship between preoperative anxiety levels and fetal cord blood TNF-α and IL-6 cytokine levels in pregnant women.

DETAILED DESCRIPTION:
This prospective observational study is planned to involve 30 volunteer patients between 18-40 years of age who will undergo elective caesarean section surgery. People with known psychiatric illness and medication use, illiterate, who do not have mental competence to understand survey questions and very urgent patients will not be included in the study.

Preoperative anxiety levels will be determined by the STAI-Continuity scale at the time of admission to the anesthesia outpatient clinic and by the STAI-State scale 1 hour before surgery.The scales will be scored as normal, mild, moderate and severe anxiety. Psychiatric consultation will be requested for patients with severe anxiety. At the end of the cesarean section, the concentration of TNF-α and IL-6 cytokines in the blood remaining from routine blood gas taken from the umbilical cord will be determined to obtain information about the state of fetal well-being.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-40 years
* Undergo elective caesarean section surgery
* Volunteer patients

Exclusion Criteria:

* People with known psychiatric illness and medication use
* Who do not have mental competence to understand survey questions
* Very urgent patients
* İlliterate

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Elective caesarean section surgery
Study Population: This prospective observational study is planned to involve 30 volunteer patients between 18-40 years of age who will undergo elective caesarean section by Obstetrics and Gynecology Department.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Correlation between preoperative anxiety level and fetal cord blood Tumor Necrosis Factor-Alfa and İnterleukin-6 cytokine levels | 1 Day
  Preoperative anxiety levels:anesthesia outpatient clinic with STAI-Continuity Scale and 1 hour before surgery with the STAI-State scale.

CONTACTS AND LOCATIONS:
Overall Officials: Yozgat Bozok University Research Hospital, Study Director — Yozgat
Locations (1):
- Yozgat Bozok University, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No